CLINICAL TRIAL: NCT01967030
Title: SWIFT: Study of Women, Infant Feeding and Type 2 Diabetes After GDM Pregnancy
Acronym: SWIFT
Status: Active, not recruiting | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Diabetes Association (Other); W.K. Kellogg Foundation (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: CN-04EGund-03-H; R01HD050625 (NIH); R01DK118409-01 (NIH); R21DK103171 (NIH); 200-2011-M-39058 (Other Grant/Funding Number: Centers for Disease Control and Prevention); R56HL148260 (NIH)
Record Dates: First submitted 2013-10-11; First posted 2013-10-22 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
Keywords: gestational diabetes mellitus; breastfeeding; obesity; type 2 diabetes; lactation; prospective; women; postpartum; incident diabetes; epidemiology; metabolomics; cardiometabolic health
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational; Breast Feeding; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We collected fasting and 2-hour post-load plasma specimens during each 2-hour 75 gram Oral Glucose Tolerance Test (OGTT) from three longitudinal research exams at 6 to 9 weeks postpartum (study baseline), and at research exams at 1 year and 2 years post-baseline. The EDTA treated plasma specimens and buffy coats are stored in cryovials at -80 degrees Centrigrade in low temperature freezers at the Division of Research Clinic in Oakland, CA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with recent GDM pregnancy: The study cohort includes women who had gestational diabetes mellitus (GDM) in their index pregnancy for study enrollment. There are two pre-defined groups: 1) women who breastfeed intensively during the first 4 months postpartum, and 2) women who mostly fed formula during the first 4 months postpartum. The study enrolled women into these pre-defined groups, but some women transitioned into mixed feeding groups after enrollment.

SUMMARY:
The overall goal of the Study of Women, Infant Feeding and Type 2 Diabetes after GDM pregnancy (SWIFT) is to determine the relation of longer and more intensive lactation, as compared to formula feeding, on progression to incident type 2 diabetes mellitus among women within several years following delivery of a GDM pregnancy. The initial study enrolled women with recent GDM at 6 to 9 weeks post-delivery to reclassify oral glucose tolerance and conduct subsequent testing of glucose tolerance to ascertain progression to overt diabetes up to two years later. Research methods were utilized to assess lactation intensity and duration quantitatively and to evaluate incidence rates of diabetes, as well as changes in blood glucose levels, insulin resistance, body weight, waist circumference, and overall adiposity from baseline and up to several years later. SWIFT is a prospective, observational cohort study of 1,035 women recruited during pregnancy who were diagnosed with gestational diabetes mellitus (GDM) via Carpenter and Coustan criteria and enrolled into the research study. We assessed the natural history of progression to prediabetes and type 2 diabetes from early postpartum for a racially and ethnically diverse cohort of women with GDM (75% minority) at high-risk for developing overt diabetes within 5-10 years post-delivery.

DETAILED DESCRIPTION:
The SWIFT study recruited women during pregnancy, and enrolled 1,035 women diagnosed with GDM who delivered a singleton, live born infant of at least 35 weeks gestation at a Kaiser Permanente Northern California hospital from 2008 to 2011, and met other study eligibility criteria. Women with recent GDM consented to three in-person research exams with the first exam at 6-9 weeks postpartum (study baseline) and the two follow up research exams continuing annually thereafter for two years post-baseline. SWIFT participants continued to be followed for clinical diagnoses of diabetes via the KPNC electronic health record system during the subsequent years through present. The study enrollment of participants began in late 2008 and ended in December 2011, and in-person follow up exams through 2014. The SWIFT cohort is racially and ethnically diverse (75% minority) with 35% Asian (1/3 South Asian, 1/3 Southeast Asian, 1/3 Chinese), 9% Black, 31% Hispanic, 23% White, and 2% mixed race/Native groups, and includes a longitudinal research Biobank, and research datasets, and clinical electronic health record data for diagnoses of diabetes and other clinical measures.

Each woman provided written informed consent for three in-person exams involving administration of the 2-hour 75 gram Oral Glucose Tolerance Test (OGTT) to reclassify glucose tolerance in women following GDM pregnancy, and numerous other research assessments. At baseline, 21 women were classified with overt diabetes and excluded from follow up, 2 women dropped out at baseline, and 2 women were ineligible. There were 1,010 women with recent GDM and no diabetes at baseline who were followed to evaluate the primary study outcome, the progression to glucose intolerance during the two year follow up period, defined as incident diabetes by American Diabetes Association (ADA) criteria from the 2-hour 75 gram OGTT glucose values, and/or clinical medical diagnosis of diabetes. The annual study follow up exams during the 2 years post-baseline occurred from 2009-2014. The study cohort continues in ongoing follow up for progression to diabetes and subsequent pregnancies via laboratory testing from the Kaiser Permanente electronic health records through present (72% remain KPNC health plan members). A 4th in person research exam is enrolling SWIFT participants in 2022-2024,

The primary exposure for the study is lactation intensity and duration assessed quantitatively using the method by Piper et al. 2001 to estimate a continuous lactation intensity and duration score up to 12 months postpartum. The study assessed infant feeding prospectively from prenatal telephone contacts to assess breastfeeding intention via a standardized method, inpatient hospital delivery records, participant infant feeding diaries, telephone contacts at 1 month postpartum, self-administered monthly mailed surveys (from 3 to 11 months postpartum), and from surveys at the three in-person annual study exams. Data collection during and after pregnancy was also obtained from electronic health records related to perinatal course (e.g., laboratory diagnosis of GDM phenotype severity: 3-hr OGTT z-score and GDM treatment, gestational age at GDM diagnosis, maternal pre-pregnancy BMI, gestational weight gain), medical history, prenatal measures, subsequent pregnancies, and the maternal and newborn outcomes.

Subsequent studies of metabolites preceding progression to overt diabetes after gestational diabetes pregnancy are underway. Investigations are ongoing to measure changes in metabolomics, proteomics and lipidomics at the baseline and follow up exams.

At each of three study exams, trained research staff assessed maternal characteristics (infant feeding, sociodemographics, medical and reproductive history, subsequent pregnancies, medication use, recurrence of GDM, physical activity, dietary intake, depression, and sleep habits/disorders), as well as breastfeeding intensity and duration, infant health, and complementary infant dietary intake using self- and interviewer-administered questionnaires. Trained research staff measured participant anthropometry and body composition via bioelectrical impedance assessment according to standardized research protocols, as well as collected, processed, and stored biospecimens from 2-hour 75 g OGTTs (fasting and 2-h plasma and buffy coat), and administered questionnaires at each in-person exam.

The SWIFT Offspring Study, an ancillary study of mother-infant dyads, conducted three in-person exams from 6-9 weeks, 6 months and 12 months to evaluate infant ponderal growth (weight and length) during the first year of life as well as sleep, infant temperament, dietary intake, skinfold thickness, breastfeeding and formula feeding, and collect saliva specimens in the infants of the SWIFT mothers.

Ongoing surveillance to ascertain new diagnoses of diabetes in the SWIFT cohort occurred both during and after the study period via the KPNC electronic health records from 2009 to 2018. The SWIFT study plans to recontact all 1,033 active participants in 2019 to conduct a fourth in-person exam at 12 years post-baseline from 2022-2024 (delayed due to COVID-19 pandemic). The fourth in-person research exam at 12-years post-baseline will reassess glucose tolerance, anthropometry, body composition and other attributes as described previously. The SWIFT study also utilizes fasting plasma specimens sampled within the early postpartum period to identify metabolites for the early prediction of future progression to type 2 diabetes. Changes in anthropometry, lifestyle behaviors, and risk factors for diabetes will also be assessed at the 12-year post-baseline in-person exam.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 45 years at delivery
* received prenatal care in Kaiser Permanente Northern California (KPNC) health care system
* Gestational Diabetes (GDM) pregnancy diagnosed using the 3-hour 100 g OGTT by Carpenter and Coustan criteria
* delivered a singleton, live birth >= 35 weeks gestation
* no pre-existing diabetes or other serious medical conditions prior to index GDM pregnancy
* no diabetes diagnosis (2-hour 75 gram OGTT) at 6 to 9 weeks postpartum for the index GDM pregnancy
* no use of thyroid medications, steroids, or other medications affecting glucose tolerance
* not planning to move from the northern California area within the subsequent 24 months
* not planning another pregnancy within the next two years
* Two infant feeding groups: women who did not lactate or did so for less than 3 weeks, OR women who provided no supplemental milk feeds at 2-4 weeks and planned to continue intensive lactation defined as <= 1 formula supplement (6 oz/day) from 6-9 weeks until 4 months or more postpartum.

Exclusion criteria:

* Women who fed both breast milk and 7-16 oz of formula (mixed feeding) during the first 4 weeks of life

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: SWIFT participants were recruited from Kaiser Permanente Northern California (KPNC) Region medical centers. Participating research field sites for the in-person research exams were located within the three primary areas:
  North area: Medical Centers in Sacramento, South Sacramento, and Roseville, and the Rancho Cordova, Elk Grove, Point West, and Folsom Medical Offices; East area: Division of Research (DOR) Research Clinic (Oakland), Hayward Medical Center and Fremont Medical Offices and Richmond Medical Center; South area: Santa Clara, and San Jose Medical Centers.
  The prospective cohort of women with GDM received prenatal care and delivered a singleton, live born infant of 35 weeks gestation or longer at a Kaiser Permanente hospital between July 2008 and October 2011.
Sampling Method: Non-Probability Sample
Enrollment: 1035 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Incident Type 2 Diabetes | baseline to 12 years postpartum
  Two-hour 75 gram oral glucose tolerance test; fasting plasma and 2-hour post-load plasma samples analyzed for glucose and insulin concentrations.

SECONDARY OUTCOMES:
Maternal weight | 2 years postpartum and 12 years post-baseline
  Body weight
Body composition | 2 years postpartum and 12 years post-baseline
  Tetra polar Bioelectrical impedance to estimate percent body fat
Maternal waist circumference | 2 years postpartum and 12 years post-baseline
  Waist circumference

OTHER OUTCOMES:
Insulin Resistance Index | 2 years postpartum and 12 years post-baseline
  Fasting plasma and 2 hour post-load plasma assayed for concentrations of glucose and insulin. These measures will be used to calculate homeostatic model assessment of insulin resistance (HOMA-IR).
Insulin secretion Index | 2 years postpartum and 12 years post-baseline
  Fasting plasma and 2 hour post-load plasma assayed for concentrations of glucose and insulin. These measures will be used to calculate the homeostatic model assessment of insulin secretion (HOMA-ß).
Metabolite profiles | Up to 12 years post-baseline
  New Ancillary Study utilizes stored fasting plasmas samples from the 3 in-person research exams in the cohort, and newly collected plasma from the 12-year follow up research exam to measure a panel of 183 targeted metabolites related to type 2 diabetes, and 1000 lipid metabolites using Mass Spectroscopy quantitative methodology. The metabolites will be measured using a panel developed by Metabolon, Inc. These metabolites will be used to identify a signature to predict progression to type 2 diabetes after Gestational diabetes pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Erica P Gunderson, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, Division of Research, Oakland, California, United States

REFERENCES:
- [Result] Gunderson EP. Impact of breastfeeding on maternal metabolism: implications for women with gestational diabetes. Curr Diab Rep. 2014 Feb;14(2):460. doi: 10.1007/s11892-013-0460-2. PMID 24402327
- [Result] Gunderson EP. The role of lactation in GDM women. Clin Obstet Gynecol. 2013 Dec;56(4):844-52. doi: 10.1097/GRF.0b013e3182a8e067. PMID 24100596
- [Result] Gunderson EP, Greenspan LC, Faith MS, Hurston SR, Quesenberry CP Jr; SWIFT Offspring Study Investigators. Breastfeeding and growth during infancy among offspring of mothers with gestational diabetes mellitus: a prospective cohort study. Pediatr Obes. 2018 Aug;13(8):492-504. doi: 10.1111/ijpo.12277. Epub 2018 Apr 24. PMID 29691992
- [Result] Batchuluun B, Al Rijjal D, Prentice KJ, Eversley JA, Burdett E, Mohan H, Bhattacharjee A, Gunderson EP, Liu Y, Wheeler MB. Elevated Medium-Chain Acylcarnitines Are Associated With Gestational Diabetes Mellitus and Early Progression to Type 2 Diabetes and Induce Pancreatic beta-Cell Dysfunction. Diabetes. 2018 May;67(5):885-897. doi: 10.2337/db17-1150. Epub 2018 Feb 7. PMID 29436377
- [Result] Davis JN, Shearrer GE, Tao W, Hurston SR, Gunderson EP. Dietary variables associated with substantial postpartum weight retention at 1-year among women with GDM pregnancy. BMC Obes. 2017 Aug 3;4:31. doi: 10.1186/s40608-017-0166-0. eCollection 2017. PMID 28794888
- [Result] Gunderson EP; Study of Women, Infant Feeding and Type 2 Diabetes After GDM Pregnancy Investigators. Lactation and Progression to Type 2 Diabetes Mellitus After Gestational Diabetes Mellitus. Ann Intern Med. 2016 Aug 16;165(4):299-300. doi: 10.7326/L16-0106. No abstract available. PMID 27538169
- [Result] Allalou A, Nalla A, Prentice KJ, Liu Y, Zhang M, Dai FF, Ning X, Osborne LR, Cox BJ, Gunderson EP, Wheeler MB. A Predictive Metabolic Signature for the Transition From Gestational Diabetes Mellitus to Type 2 Diabetes. Diabetes. 2016 Sep;65(9):2529-39. doi: 10.2337/db15-1720. Epub 2016 Jun 23. PMID 27338739
- [Result] Gunderson EP, Hurston SR, Ning X, Lo JC, Crites Y, Walton D, Dewey KG, Azevedo RA, Young S, Fox G, Elmasian CC, Salvador N, Lum M, Sternfeld B, Quesenberry CP Jr; Study of Women, Infant Feeding and Type 2 Diabetes After GDM Pregnancy Investigators. Lactation and Progression to Type 2 Diabetes Mellitus After Gestational Diabetes Mellitus: A Prospective Cohort Study. Ann Intern Med. 2015 Dec 15;163(12):889-98. doi: 10.7326/M15-0807. Epub 2015 Nov 24. PMID 26595611
- [Result] Gunderson EP, Hurston SR, Dewey KG, Faith MS, Charvat-Aguilar N, Khoury VC, Nguyen VT, Quesenberry CP Jr. The study of women, infant feeding and type 2 diabetes after GDM pregnancy and growth of their offspring (SWIFT Offspring study): prospective design, methodology and baseline characteristics. BMC Pregnancy Childbirth. 2015 Jul 17;15:150. doi: 10.1186/s12884-015-0587-z. PMID 26177722
- [Result] Gunderson EP, Kim C, Quesenberry CP Jr, Marcovina S, Walton D, Azevedo RA, Fox G, Elmasian C, Young S, Salvador N, Lum M, Crites Y, Lo JC, Ning X, Dewey KG. Lactation intensity and fasting plasma lipids, lipoproteins, non-esterified free fatty acids, leptin and adiponectin in postpartum women with recent gestational diabetes mellitus: the SWIFT cohort. Metabolism. 2014 Jul;63(7):941-50. doi: 10.1016/j.metabol.2014.04.006. Epub 2014 Apr 13. PMID 24931281
- [Result] Gunderson EP, Crites Y, Chiang V, Walton D, Azevedo RA, Fox G, Elmasian C, Young S, Salvador N, Lum M, Hedderson MM, Quesenberry CP, Lo JC, Ferrara A, Sternfeld B. Influence of breastfeeding during the postpartum oral glucose tolerance test on plasma glucose and insulin. Obstet Gynecol. 2012 Jul;120(1):136-43. doi: 10.1097/AOG.0b013e31825b993d. PMID 22914402
- [Result] Gunderson EP, Hedderson MM, Chiang V, Crites Y, Walton D, Azevedo RA, Fox G, Elmasian C, Young S, Salvador N, Lum M, Quesenberry CP, Lo JC, Sternfeld B, Ferrara A, Selby JV. Lactation intensity and postpartum maternal glucose tolerance and insulin resistance in women with recent GDM: the SWIFT cohort. Diabetes Care. 2012 Jan;35(1):50-6. doi: 10.2337/dc11-1409. Epub 2011 Oct 19. PMID 22011407
- [Result] Gunderson EP, Matias SL, Hurston SR, Dewey KG, Ferrara A, Quesenberry CP Jr, Lo JC, Sternfeld B, Selby JV. Study of Women, Infant Feeding, and Type 2 diabetes mellitus after GDM pregnancy (SWIFT), a prospective cohort study: methodology and design. BMC Public Health. 2011 Dec 23;11:952. doi: 10.1186/1471-2458-11-952. PMID 22196129
- [Result] Gunderson EP, Jaffe MG. Pregnancy and Subsequent Glucose Intolerance in Women of Childbearing Age: Heeding the Early Warning Signs for Primary Prevention of Cardiovascular Disease in Women. JAMA Intern Med. 2017 Dec 1;177(12):1742-1744. doi: 10.1001/jamainternmed.2017.4768. No abstract available. PMID 29049465
- [Result] Khan SR, Mohan H, Liu Y, Batchuluun B, Gohil H, Al Rijjal D, Manialawy Y, Cox BJ, Gunderson EP, Wheeler MB. The discovery of novel predictive biomarkers and early-stage pathophysiology for the transition from gestational diabetes to type 2 diabetes. Diabetologia. 2019 Apr;62(4):687-703. doi: 10.1007/s00125-018-4800-2. Epub 2019 Jan 15. PMID 30645667
- [Result] Faith MS, Hittner JB, Hurston SR, Yin J, Greenspan LC, Quesenberry CP Jr, Gunderson EP; SWIFT Offspring Study Investigators. Association of Infant Temperament With Subsequent Obesity in Young Children of Mothers With Gestational Diabetes Mellitus. JAMA Pediatr. 2019 May 1;173(5):424-433. doi: 10.1001/jamapediatrics.2018.5199. PMID 30855657
- [Result] Lai M, Liu Y, Ronnett GV, Wu A, Cox BJ, Dai FF, Rost HL, Gunderson EP, Wheeler MB. Amino acid and lipid metabolism in post-gestational diabetes and progression to type 2 diabetes: A metabolic profiling study. PLoS Med. 2020 May 20;17(5):e1003112. doi: 10.1371/journal.pmed.1003112. eCollection 2020 May. PMID 32433647
- [Result] Lai M, Al Rijjal D, Rost HL, Dai FF, Gunderson EP, Wheeler MB. Underlying dyslipidemia postpartum in women with a recent GDM pregnancy who develop type 2 diabetes. Elife. 2020 Aug 4;9:e59153. doi: 10.7554/eLife.59153. PMID 32748787
- [Result] Vandyousefi S, Davis JN, Gunderson EP. Association of infant diet with subsequent obesity at 2-5 years among children exposed to gestational diabetes: the SWIFT study. Diabetologia. 2021 May;64(5):1121-1132. doi: 10.1007/s00125-020-05379-y. Epub 2021 Jan 26. PMID 33495846
- [Result] Zhang Z, Lai M, Piro AL, Alexeeff SE, Allalou A, Rost HL, Dai FF, Wheeler MB, Gunderson EP. Intensive lactation among women with recent gestational diabetes significantly alters the early postpartum circulating lipid profile: the SWIFT study. BMC Med. 2021 Oct 8;19(1):241. doi: 10.1186/s12916-021-02095-1. PMID 34620173
- [Result] Zhang Z, Piro AL, Allalou A, Alexeeff SE, Dai FF, Gunderson EP, Wheeler MB. Prolactin and Maternal Metabolism in Women With a Recent GDM Pregnancy and Links to Future T2D: The SWIFT Study. J Clin Endocrinol Metab. 2022 Aug 18;107(9):2652-2665. doi: 10.1210/clinem/dgac346. PMID 35666146
- [Result] Khan SR, Manialawy Y, Obersterescu A, Cox BJ, Gunderson EP, Wheeler MB. Diminished Sphingolipid Metabolism, a Hallmark of Future Type 2 Diabetes Pathogenesis, Is Linked to Pancreatic beta Cell Dysfunction. iScience. 2020 Sep 15;23(10):101566. doi: 10.1016/j.isci.2020.101566. eCollection 2020 Oct 23. PMID 33103069
- [Result] Matias SL, Dewey KG, Quesenberry CP Jr, Gunderson EP. Maternal prepregnancy obesity and insulin treatment during pregnancy are independently associated with delayed lactogenesis in women with recent gestational diabetes mellitus. Am J Clin Nutr. 2014 Jan;99(1):115-21. doi: 10.3945/ajcn.113.073049. Epub 2013 Nov 6. PMID 24196401
- See also: Breastfeeding Research conducted at the KPNC, Division of Research, Oakland CA — https://divisionofresearch.kaiserpermanente.org/researchers/gunderson-erica
- See also: BMJ Summarizes the Primary Findings from the SWIFT Study 2015 — https://www.bmj.com/content/351/bmj.h6255
- See also: SWIFT Study Website — http://www.kp.org/swiftstudy